CLINICAL TRIAL: NCT03059160
Title: Open Label Trial of Triheptanoin (UX007) in Treatment of Rett Syndrome.
Acronym: UX007
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Principal Investigator, Prof. Bruria Ben-Zeev MD, Head of pediatric neurology unit, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3027-16-SMC
Record Dates: First submitted 2017-02-02; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Rett Syndrome
Keywords: Rett syndrome, Triheptanoic acid, Walking, EEG
MeSH Terms: conditions — Rett Syndrome | interventions — triheptanoin

STUDY DESIGN:
Intervention Model Description: open label study with one doze
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- open label (Experimental)
  Interventions: Drug: Tridecanoic Acid

INTERVENTIONS:
Drug: Tridecanoic Acid — 3 times daily oral doze of the drug for 20 weeks with 4 weeks of baseline and 4 weeks of washout
  Other Names: triheptanoin

SUMMARY:
This is a single-center, exploratory, open-label study in 10 girls diagnosed with Rett Syndrome. The study will consist of the following 4 parts: Screening/Baseline run-in, Titration/Dose-Setting, Treatment, and Washout/Follow-up.

DETAILED DESCRIPTION:
1. Screening and baseline assessments (4 weeks before first treatment): After having the parents sign an informed consent, eligible patients will undergo baseline assessments (safety and disease variables) as follows:

   * Physical examination
   * Vital signs: sitting Blood Presure (BP),Heart Rate (HR) and respiratory rate, arm pit temperature.
   * Baseline height and weight parameters
   * ECG (ElectroCardioGraphy)
   * 3-hour video EEG (ElectroEncephaloGram)
   * 24-hour NOX-T3 (Portable Sleep Monitor) recording
   * QOL (Quality of Life) and Rett Syndrome-specific functional/severity questionnaires
   * Laboratory blood tests, including endocrinology, hematology, and biochemistry.
   * Parents will be requested to fill in a diary and record on a daily basis seizure occurrence for at least 4 weeks before first treatment. In addition they will be asked to record their top 3 concerns pertaining to the care and overall well-being of the patient.
2. Treatment period (20 weeks):

   1. Initial and final dose setting (2 weeks): UX007 will be titrated in each patient over 2 weeks to a dose of 1-4 grams per kilogram per day (based on age). If a subject cannot tolerate titrating up to the 1-4 g/kg/day dose level, the dose should be titrated to the maximum tolerated dose as determined by the Investigator. At the end of the Titration Period, the subject will be maintained on the maximum UX007 dose achieved during the Titration Period for the duration of the study.

      The following assessments will be performed:

      • QOL and RTT-specific functional/severity questionnaires
   2. Final dose (18 weeks): Patients will receive a dose of UX007 as determined in the Titration/Dose Setting period. They will be followed up by the Investigator and undergo safety and disease-related assessments as follows (schedules outlined in the protocol):

      * Physical examination
      * Vital signs (sitting BP, HR and respiratory rate, oral temperature)
      * Height and weight parameters
      * ECG
      * 3-hour video EEG
      * 24-hour NOX recording
      * Motor assessment
      * QOL and RTT-specific functional/severity questionnaires
      * Laboratory blood tests, including endocrinology, hematology, and biochemistry.
      * Data collection from parents' diaries

4. Post-Washout Follow-up/End-of-Study:

Within approximately six (6) weeks after last dose administration, a termination visit will be scheduled. The following activities will take place:

* Physical examination
* Vital signs (sitting BP, HR and respiratory rate, oral temperature)
* Height and weight parameters
* ECG
* 3-hour video EEG
* 24-hour NOX recording
* Motor assessment
* QOL and RTT-specific functional/severity questionnaires
* Laboratory blood tests, including endocrinology, hematology, and biochemistry.
* Data collection from parent's diaries
* Decision regarding continued administration of UX007 to patients who benefitted from the trial after the dechallenge period

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 5 to18 years (inclusive).
* A classical diagnosis of RTT, defined according to the internationally agreed 2010 Rett Search criteria, and with MECP2 pathogenic mutation.
* Patients with one or both of the following:

  * At least 2 seizures per month as per history during the four-week baseline period according to parent diary or per 3 hours video EEG recording
  * Walking abilities, independent or with support
* Patients with breathing abnormalities as recorded by baseline NOX recording.

Exclusion Criteria:

* Patients with significant metabolic, liver, cardiac, or respiratory morbidity not related to RTT
* Patients with significant liver, cardiac or respiratory morbidity related to RTT

Ages: 5 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 10 (Estimated)
Dates: Start 2017-04-01 (Estimated); Primary Completion 2018-04-01 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
The number of patients with adverse events. | 30 weeks
  The number of patients which will show adverse events during the screening, treatment and washout periods.
The number of patients with ECG changes | 30 weeks
  The number of patients that show ECG changes and the type of change during the screening, treatment and washout periods.
The number of patients with changes in vital signs. | 30 weeks
  The number of patients which will show change in vital signs during the screening, treatment and washout periods including bloodpressure, heart rate, respiration rate and body temperature.
The number of patients with changes in physical examination. | 30 weeks
  The number of patients who show a change in their physical examination during the screening, treatment and washout periods including height, neurological findings, change in size of liver and spleen , skin changes.
The number of patients with changes in BMI | 30 weeks
  The number of patients who will show change in BMI and its direction during the screening, treatment and washout periods.
The number of patients with changes in laboratory examination including hematology, biochemistry and endocrinological measurements | 30 weeks
  The number of patients who will show changes in laboratory examination including hematology, biochemistry and endocrinological measurements during the screening, treatment and washout periods.

SECONDARY OUTCOMES:
Change in seizure frequency during treatment with triheptanoin in Rett syndrome | 30 weeks
  The change in number of seizures in each patient from the base line period to the treatment period and washout period

CONTACTS AND LOCATIONS:
Overall Officials: Bruria Ben-Zeev, MD, Principal Investigator — Head of pediatric neurology unit in Sheba medical center

IPD SHARING:
Plan to Share IPD: Yes
the final results of the study will be shared with ultragenix pharmaceutical and with other RETT syndrome researchers